CLINICAL TRIAL: NCT03778073
Title: A Phase 1 Study of Cosibelimab (TG-1501) in Subjects With Relapsed or Refractory Lymphoma
Brief Title: Study of Cosibelimab in Subjects With Relapsed or Refractory Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic/Business Decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-1501-101
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: B-cell Non Hodgkin Lymphoma; Richter's Transformation
Keywords: relapsed or refractory
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence | interventions — ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Cosibelimab (TG-1501) single-agent
  Interventions: Drug: Cosibelimab
- Cohort B (Experimental): Cosibelimab + Ublituximab + Bendamustine combination
  Interventions: Drug: Cosibelimab + Ublituximab + Bendamustine combination
- Cohort C (Experimental): Cosibelimab + Ublituximab + Bendamustine combination
  Interventions: Drug: Cosibelimab + Ublituximab + Bendamustine combination

INTERVENTIONS:
Drug: Cosibelimab — Intravenous infusion on Days 1 and 15 of every 28-day cycle or only on Day 1 of every 28-day cycle
  Arms: Cohort A
Drug: Cosibelimab + Ublituximab + Bendamustine combination — Cosibelimab (Intravenous infusion):
  Cycle 1-6 Days 1&15, Cycles 7-12 Day 1, Cycles 15-24 Day 1 every 3 cycles;
  Ublituximab (Intravenous infusion):
  Cycles 1-6 Day 1, Cycles 9-24 every 3 Cycles;
  Bendamustine (Intravenous infusion):
  Cycle 1 Days 2&3, Cycles 2-6 Days 1&2.
  Arms: Cohort B
Drug: Cosibelimab + Ublituximab + Bendamustine combination — Cosibelimab (Intravenous infusion):
  Cycle 1-12 Day 1, Cycles 15-24 Day 1 every 3 cycles;
  Ublituximab (Intravenous infusion):
  Cycles 1-6 Day 1, Cycles 9-24 every 3 Cycles;
  Bendamustine (Intravenous infusion):
  Cycle 1 Days 2&3, Cycles 2-6 Days 1&2.
  Arms: Cohort C

SUMMARY:
Phase 1 open label, multi-center, dose-escalation study for individuals with relapsed or refractory B-cell Non Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
This study will evaluate the safety profile, pharmacokinetics, and efficacy of single-agent cosibelimab as well as the combination of Cosibelimab + Ublituximab + Bendamustin.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed relapsed or refractory B-cell non-Hodgkin lymphoma (NHL).
* Measurable disease and adequate organ function as specified in the protocol

Key Exclusion Criteria:

* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or prior therapy with bendamustine.
* Subjects receiving cancer therapy or investigational drug within 21 days of Cycle 1 Day 1.
* Prior autologous stem cell transplant within 3 months
* Active Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events That Are Related to Treatment | 6 months of therapy
  Number of Participants With Treatment-Related Adverse Events, any potential abnormal laboratory results and any dose-limiting toxicities

SECONDARY OUTCOMES:
Overall Response Rate | Up to 12 months
  Objective response in subjects treated with interventions

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Tucson, Arizona
  - TG Therapeutics Investigational Trial Site, Fayetteville, Arkansas
  - TG Therapeutics Investigational Trial Site, Peoria, Illinois
  - TG Therapeutics Investigational Trial Site, Fort Wayne, Indiana
  - TG Therapeutics Investigational Trial Site, Fairway, Kansas
  - TG Therapeutics Investigational Trial Site, Louisville, Kentucky
  - TG Therapeutics Investigational Trial Site, Charlotte, North Carolina
  - TG Therapeutics Investigational Trial Site, Seattle, Washington